CLINICAL TRIAL: NCT07030426
Title: A Multi-center, Randomized, Open-label, Parallel-group, Feasibility-controlled Trial of Vaginal Estrogen for Improvement of Outcomes Following Pelvic Organ Prolapse Surgery
Brief Title: Vaginal Estrogen for Improvement of Outcomes Following Pelvic Organ Prolapse Surgery
Acronym: VEPO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Sarah Wozney, Assistant Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ref: No 70577
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Organ Prolapse (POP)
Keywords: pelvic organ prolapse; vaginal estrogen; pelvic organ prolapse surgery; pelvic organ prolapse repair
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Vaginal Estrogen Group (No Intervention): No vaginal estrogen
- Twice Weekly Vaginal Estrogen Group (Active Comparator): Twice Weekly Vaginal Estrogen
  Interventions: Drug: Vaginal Estrogen - Twice Weekly
- Daily Vaginal Estrogen Group (Active Comparator): Daily Vaginal Estrogen
  Interventions: Drug: Vaginal Estrogen - Daily

INTERVENTIONS:
Drug: Vaginal Estrogen - Twice Weekly — Twice weekly for six weeks following pelvic organ prolapse repair surgery. 0.5 grams of cream per vagina at bedtime .
  Other Names: Conjugated Estrogens CSD, 0.625 mg/g, Vaginal Cream
  Arms: Twice Weekly Vaginal Estrogen Group
Drug: Vaginal Estrogen - Daily — Daily for six weeks following pelvic organ prolapse repair surgery. 0.5 grams of cream per vagina at bedtime.
  Other Names: Conjugated Estrogens CSD, 0.625 mg/g, Vaginal Cream
  Arms: Daily Vaginal Estrogen Group

SUMMARY:
This open-label randomized control trial will study the use of vaginal estrogen in the first six weeks after pelvic organ prolapse (POP) repair surgery. This is a pilot trial that will examine the feasibility of the study, focussing on recruitment rates. Participants will be randomized to one of three groups; (1) no vaginal estrogen for 6 weeks, (2) vaginal estrogen twice weekly for 6 weeks, or (3) vaginal estrogen daily for 6 weeks. Participants will be seen at 6 weeks post surgery, 6 months post surgery, 1 year and 2 years post surgery. Additional outcomes will include patient satisfaction, Genitourinary Syndrome of Menopause (GSM) symptoms, post-operative complications, adherence and safety.

DETAILED DESCRIPTION:
Multi-center, randomized, open-label, parallel-group, feasibility-controlled trial

The intervention is the use of vaginal estrogen for 6 weeks after pelvic organ prolapse surgery. Participants will be randomized into 3 groups:

1. No vaginal estrogen
2. Vaginal estrogen 2 times per week
3. Vaginal estrogen daily

Participants may be enrolled after diagnosis of pelvic organ prolapse and decision to proceed with surgery. Participants will be seen for a randomization visit within 6 weeks of their scheduled surgery. The intervention lasts from the day of surgery until 6 weeks after surgery. Participants will be seen for a post-operative follow-up visit at 6 weeks, and study follow-up visits at 6 months, 1 year and 2 years.

Sample Size: N=60 in each group, for a total of N=180 participants. For this pilot trial, we will recruit approximately 15% of the sample size required for the full-scale trial. Data from this pilot trial will be used to adjust the event rate in the sample size calculation for the full trial, if needed. Our sample size accounts for a non-compliance rate of 5% and a loss to follow-up rate of 5%.

After enrollment, participants will complete a baseline questionnaire that collects information on demographics and health history. This may be completed online via an email link sent through REDCap, in person on a hard copy questionnaire, or the questions can be administered verbally by study staff.

After enrollment, a study investigator or delegate will complete a case report for that collects additional information on the participant's pregnancy and pelvic health history.

At each study visit, a study investigator or delegate will complete a case report form that captures any changes in the participant's health history since the previous visit.

At all post-surgical visits, a study investigator or delegate will collect information in these same case report forms on complications and treatment failure. The questions in these case report forms will be administered verbally, with verification through chart review as appropriate or as needed.

At each study visit a Pelvic Organ Prolapse Quantification (POP-Q) and Visual Analog Scale (VAS) on GSM symptoms assessment will be completed by a study investigator or medical learner under direct supervision of a study investigator. As well, height, weight and blood pressure will be measured. If any of these are collected/done for clinical reasons at the same visit, the clinically collected data will be used for study purposes. The measurements and assessments will not be repeated for study purposes.

At each study visit the Prolapse Quality of Life Questionnaire (P-QOL) and incontinence questionnaires including the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF), the Incontinence Impact Questionnaire Short Form (IIQ-7), and the Urogenital Distress Inventory Short Form (UDI-6) will be administered. These may be completed online via an email link sent through REDCap, in person on a hard copy questionnaire, or the questions can be administered verbally by study staff.

At the 6 week and 6 month post-surgical visit the Surgical Satisfaction Questionnaire (SSQ-8) will be administered. These may be completed online via an email link sent through REDCap, in person on a hard copy questionnaire, or the questions can be administered verbally by study staff.

At the 6 week post-surgical visit adherence to the study intervention will be assessed through collection of study product diaries and by querying participants on vaginal estrogen usage in the intervention period.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all the following inclusion criteria to be eligible for enrollment into the study:

1. Participant who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
2. The participant has given written consent after the study has been explained according to local regulatory requirements and before any study specific procedures.
3. Age ≥18 years at the time of consent.
4. Undergoing an apical suspension (vaginal or abdominal, mesh or native tissue) for pelvic organ prolapse at one of the participating centers.
5. Primary or recurrent prolapse surgery without a history of mesh surgery.
6. Willing to complete surveys related to demographics, pelvic health and function, and sexual health and function.
7. Plans to reside in the study area for at least 2 years after their surgery.

Exclusion Criteria

Any individual meeting any of the following criteria is not eligible for participation in this study:

1. Participant undergoing anterior and/or posterior repair only (no apical prolapse repair).
2. Participant undergoing obliterative procedures.
3. Participant with a history of mesh surgery for prolapse.
4. Participant undergoing uterine sparing surgery.
5. Participant with a contraindication to vaginal estrogen use, including but not limited to the following list, at the discretion of the study investigator:

   * Patients who are hypersensitive to the drug or to any ingredient in the formulation or component of the container.
   * Liver dysfunction or disease as long as liver function tests have failed to return to normal.
   * Known or suspected estrogen-dependent malignant neoplasia (e.g. endometrial cancer).
   * Endometrial hyperplasia.
   * Known, suspected, or past history of breast cancer.
   * Undiagnosed abnormal genital bleeding.
   * Known or suspected pregnancy
   * Active or past history of arterial thromboembolic disease (e.g. stroke, myocardial infarction, coronary heart disease).
   * Partial or complete loss of vision due to ophthalmic vascular disease.
   * Known thrombophilic disorders (e.g., protein C, protein S OR antithrombin deficiency); prothrombin mutation or anticardiolipin antibodies).
6. Any conditions that, in the Investigator's judgement, may interfere with participant's ability to comply with study procedures or receipt of care, such as behavioral or cognitive impairment or neuropsychiatric illness.
7. Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 12 months
  For the primary feasibility outcome, the trial will be considered feasible if at least 75% of the target sample can be recruited in 12 months.

SECONDARY OUTCOMES:
Loss to Follow Up Rate - 6 months | 6 Months post surgery
  Loss to follow up rates at each of the study end points measured as n/N (%).
Loss to Follow Up Rate - 1 year | 1 year post surgery
  Loss to follow up rates at each of the study end points measured as n/N (%).
Loss to Follow Up Rate - 2 years | 2 years post surgery
  Loss to follow up rates at each of the study end points measured as n/N (%).
Patient Satisfaction - 6 weeks | 6 weeks post surgery
  Patient satisfaction will be assessed using the Surgical Satisfaction Questionnaire (SSQ-8). This questionnaire measures satisfaction with the surgical procedure on a scale from 8 (most satisfied) to 40 (least satisfied).
Patient Satisfaction - 6 months | 6 months post surgery
  Patient satisfaction will be assessed using the Surgical Satisfaction Questionnaire (SSQ-8). This questionnaire measures satisfaction with the surgical procedure on a scale from 8 (most satisfied) to 40 (least satisfied).
GSM Symptoms - 6 weeks | 6 weeks post surgery
  GSM symptoms will be assessed using the Visual Analog Scale (VAS) on GSM symptoms. It assesses 5 symptoms (dryness, itching, burning, dyspareunia, and dysuria) on a scale from 0 - 10, from no symptoms to severe symptoms.
GSM Symptoms - 6 months | 6 weeks post surgery
  GSM symptoms will be assessed using the Visual Analog Scale (VAS) on GSM symptoms. It assesses 5 symptoms (dryness, itching, burning, dyspareunia, and dysuria) on a scale from 0 - 10, from no symptoms to severe symptoms.
GSM Symptoms - 1 year | 1 year post surgery
  GSM symptoms will be assessed using the Visual Analog Scale (VAS) on GSM symptoms. It assesses 5 symptoms (dryness, itching, burning, dyspareunia, and dysuria) on a scale from 0 - 10, from no symptoms to severe symptoms.
GSM Symptoms - 2 years | 2 years post surgery
  GSM symptoms will be assessed using the Visual Analog Scale (VAS) on GSM symptoms. It assesses 5 symptoms (dryness, itching, burning, dyspareunia, and dysuria) on a scale from 0 - 10, from no symptoms to severe symptoms.
Prolapse Quality of Life - 6 weeks | 6 weeks post surgery
  The impact of pelvic organ prolapse on the participant's quality of life will be assessed using the Prolapse Quality of Life Questionnaire (P-QOL). The P-QOL questionnaire is a self-reported tool that contains 20 questions representing nine quality of life domains: general health, prolapse impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy and severity measures. Scores in each domain range from 0 to 100. Higher scores indicate a greater impairment of quality of life, and lower scores indicate a good quality of life.
Prolapse Quality of Life - 6 months | 6 months post surgery
  The impact of pelvic organ prolapse on the participant's quality of life will be assessed using the Prolapse Quality of Life Questionnaire (P-QOL). The P-QOL questionnaire is a self-reported tool that contains 20 questions representing nine quality of life domains: general health, prolapse impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy and severity measures. Scores in each domain range from 0 to 100. Higher scores indicate a greater impairment of quality of life, and lower scores indicate a good quality of life.
Prolapse Quality of Life - 1 year | 1 year post surgery
  The impact of pelvic organ prolapse on the participant's quality of life will be assessed using the Prolapse Quality of Life Questionnaire (P-QOL). The P-QOL questionnaire is a self-reported tool that contains 20 questions representing nine quality of life domains: general health, prolapse impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy and severity measures. Scores in each domain range from 0 to 100. Higher scores indicate a greater impairment of quality of life, and lower scores indicate a good quality of life.
Prolapse Quality of Life - 2 years | 2 years post surgery
  The impact of pelvic organ prolapse on the participant's quality of life will be assessed using the Prolapse Quality of Life Questionnaire (P-QOL). The P-QOL questionnaire is a self-reported tool that contains 20 questions representing nine quality of life domains: general health, prolapse impact, role limitations, physical limitations, social limitations, personal relationships, emotions, sleep/energy and severity measures. Scores in each domain range from 0 to 100. Higher scores indicate a greater impairment of quality of life, and lower scores indicate a good quality of life.
Complications - 6 weeks | 6 weeks post surgery
  A composite measure of the incidence of mesh erosion, urinary tract and/or surgical site infections and treatment failure.
Complications - 6 months | 6 months post surgery
  A composite measure of the incidence of mesh erosion, urinary tract and/or surgical site infections and treatment failure.
Treatment Failure - 1 year | 1 year post surgery
  A composite measure of the incidence of mesh erosion and treatment failure.
Treatment Failure - 2 years | 2 years post surgery
  A composite measure of the incidence of mesh erosion and treatment failure.

OTHER OUTCOMES:
Adherence | 6 weeks post surgery
  Adherence rates during the 6-week intervention period based on groups assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Wozney, MD, MScHQ, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - Kingston Health Sciences Centre, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The de-identified study data in the REDCap database will be retained on the Queen's CAC system for 15 years after study results are published. After the 15 year data retention period the data and data dictionary from the study REDCap database will be made available in a public data archive such as the Queen's University Library Research Data Archive in the Scholars Portal Dataverse.
Supporting Information: Study Protocol, ICF
Time Frame: 15 years after the study results are published.
Access Criteria: The data and data dictionary from the study REDCap database will be made available in a public data archive such as the Queen's University Library Research Data Archive in the Scholars Portal Dataverse.